CLINICAL TRIAL: NCT01918930
Title: A Tissue Procurement and Examination Substudy of Study CP-MGA271-01 (NCT01391143)
Brief Title: Tissue Procurement Substudy for Participants in Study CP-MGA271-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to accrue as planned for optional biopsies
Sponsor: MacroGenics (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP-MGA271-01a
Record Dates: First submitted 2013-07-30; First posted 2013-08-08 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Melanoma
Keywords: Melanoma; Accessible tumors; B7-H3 positive tumors
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGA271 (Experimental): MGA271 (administered in main study CP-MGA271-01)
  Interventions: Biological: MGA271

INTERVENTIONS:
Biological: MGA271 — MGA271 anti-B7-H3 monoclonal antibody

SUMMARY:
The purpose of this study is to gain a better understanding about how the study drug MGA271 works. No test drug will be given in this study. Patients with easily accessible tumors at the screening visit for participation in Study CP-MGA271-01 will be asked to participate in this substudy. Patients will undergo two excisional biopsies, punch biopsies, or core needle biopsies.

DETAILED DESCRIPTION:
Patients with easily accessible tumors (generally, metastatic deposits involving skin, subcutaneous tissues, or peripheral lymph node whose excision would not require general anaesthesia or the invasion of a body cavity) at the screening visit for participation in Study CP-MGA271-01 (the main study) will be asked to participate in this substudy. After providing appropriate informed consent, patients will undergo excisional biopsy, punch biopsy, or core needle biopsy of the accessible tumor prior to receiving study drug in the main study and then again after the first cycle of study drug is completed.

Some of the biopsy tissue will be sent to a central laboratory for research purposes. The central lab will analyze the tissue to see what effects that the study drug might have on tumors.

ELIGIBILITY:
Inclusion Criteria:

* Qualified, by meeting all inclusion and exclusion criteria, for participation in Study CP-MGA271-01.
* Must have provided informed consent to participate in Study CP-MGA271-01.
* Must have accessible tumors (generally speaking, metastatic deposits involving skin, subcutaneous tissue, or peripheral lymph node whose excision, punch biopsy, or core needle biopsy would not require general anaesthesia or the invasion of a body cavity).
* Willing to undergo two minor surgical procedures with no expectation of personal benefit
* Have provided Informed Consent for this substudy as indicated by a signature on an approved consent document obtained from the patient or his/her legally authorized representative

Exclusion Criteria:

* Any medical condition that would contraindicate the use of local or locoregional anaesthesia, or conscious sedation for the intended minor surgical procedure.
* Any medical condition (eg. skin disease or bleeding diathesis) that would hinder wound healing following a minor surgical procedure.
* Dementia or altered mental status that would preclude understanding and rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mechanism of Action | up to 50 days
  Exploratory analyses from immunohistochemistry (IHC) and flow cytometry testing to determine the effect of MGA271 on tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — MacroGenics
Locations (7):
- United States (7):
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Hospital of the University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No